CLINICAL TRIAL: NCT05934877
Title: Optimizing PrEP Implementation and Cost-effectiveness Among Sexual and Gender Minority Individuals With a Substance Use Disorder
Brief Title: ASK-PrEP (Assistance Services Knowledge-PrEP)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: President Trump's Executive Order
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: Weill Medical College of Cornell University (Other); University of California, Los Angeles (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: R01DA056888 (NIH)
Record Dates: First submitted 2023-05-23; First posted 2023-07-07 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-05

CONDITIONS: Substance Use Disorders; HIV
Keywords: PrEP; HIV; MSM; transgender women; substance use disorder
MeSH Terms: conditions — Substance-Related Disorders | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Two randomly assigned arms (3:1) into ASK-PrEP Stepped Care (PrEP navigation) or Standard of Care (SOC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASK-PrEP (Experimental): ASK-PrEP is a 5-session PrEP navigation intervention, with text-messaging support, to advance through the PrEP Care Continuum by identifying the individual needs and barriers to PrEP care, including substance use and behavioral health needs; adherence goal(s); and methods to achieve adherence.
  Intervention/treatment: PrEP navigation + text messaging Participants receive 5 PrEP navigation sessions within 3 months plus a weekly culturally specific, scripted text message. Participants that do not respond to the ASK-PrEP intervention at the 3-month assessment are re-randomized (1:1) and stepped up to receive ASK-PrEP plus CM or CM alone.
  Interventions: Behavioral: PrEP navigation + text messaging; Behavioral: Contingency Management
- Education and Information (Experimental): The Standard of Care (SOC) intervention includes a 20-30-minute session of PrEP information and where to access PrEP in Los Angeles. The same session is repeated at the 3-month assessment.
  Participants randomized to the SOC arm receive 2 educational/informational sessions on PrEP misconceptions, uptake, and adherence. The sessions occur at baseline and the 3-month assessment.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: PrEP navigation + text messaging — Using a client-centered approach, the PrEP navigator works to link participants into SUD treatment and other ancillary behavioral health and support services, according to their unique barriers, with the ultimate goal of PrEP initiation, adherence, and persistence; services may include mental healthcare, counseling for intimate partner violence, food insecurity, housing instability, hormone therapy. Text-messaging support includes once weekly text message.
  Arms: ASK-PrEP
Behavioral: Standard of Care — The SOC arm provides PrEP education, information, and referrals. Those randomized to the SOC arm receive an approximate 20-30-minute educational session on PrEP, and will be given a PrEP pamphlet and list of clinics that provide PrEP in LAC.
  Arms: Education and Information
Behavioral: Contingency Management — Non-responders in the ASK-PrEP arm will be stepped and re-randomized (1:1) to Contingency Management (CM), either in concert with ASK-PrEP or alone. CM is a progressive contingency schedule. Participants submit a thrice weekly urine sample. Participants will receive a voucher-based escalating reinforcement schedule. Successive urine samples that are nonreactive for the metabolites of their identified SUD will escalate their voucher point value. Each three consecutive nonreactive urine samples will receive bonus voucher points. A reactive urine sample will place the participant at the initial voucher point value; however, a rapid reset procedure allows participants to return to their place in the escalating schedule following three consecutive nonreactive urine samples. Voucher points can be redeemed at any time during the study for goods or services that promote a pro-social and healthy lifestyle.
  Arms: ASK-PrEP

SUMMARY:
ASK-PrEP is a two-arm randomized controlled trial (RCT), with a Stepped Care approach, among HIV-negative trans women and men who have sex with men with a substance use disorder (SUD). Participants will be randomized (3:1) to the ASK-PrEP Stepped Care arm or Standard of Care (SOC). Participants in the ASK-PrEP Stepped Care arm will receive 5 PrEP navigation sessions, with weekly text-messaging support, delivered over 3 months, at which point they will be assessed for intervention response. Responders will be maintained for an additional 3 months in ASK-PrEP to receive an additional 5 PrEP navigation session with weekly text-messaging support, while non-responders will receive added attention to their SUD via contingency management (CM). Non-responders will be re-randomized (1:1) to either a) receive ASK-PrEP + CM, or b) shift the primary focus to their SUD (CM alone) for an additional 3 months.

DETAILED DESCRIPTION:
ASK-PrEP is a two-arm randomized controlled trial (RCT), with a Stepped Care approach, to determine the optimal (considering effectiveness and cost-effectiveness) intervention, or combined interventions for advancement along the PrEP Care Continuum, and reductions in substance use among HIV-negative trans women (TW) and men who have sex with me (MSM), with a substance use disorder (SUD; N=250). After screening, informed consent, and baseline assessment, participants will be randomized (3:1) into one of two arms: ASK-PrEP Stepped Care or Standard of Care (SOC) control. At 3-month follow-up assessments, responders will be maintained in ASK-PrEP for an additional 3 months; non-responders will be stepped up and re-randomized (1:1) to either ASK-PrEP+CM or CM alone. Thus, non-responders will receive added attention to their SUD via CM; i.e., non-responders will either: a) receive CM in addition to a continued focus on PrEP adherence and other behavioral health issues (ASK-PrEP+CM), or b) shift the primary attention to their SUD (CM alone). Participants may choose to initiate daily oral PrEP (Truvada or Descovy) or long-acting injectable Cabotegravir. The 3-month step criteria are based on: 1) PrEP initiation and adherence; 2) substance use; and 3) HIV sexual risk behaviors if the participant has not initiated PrEP. The study uses repeated assessments at baseline and at 3-, 6-, 9-, and 12-months post-enrollment, via an "intent-to-treat" design, where all assessments are administered to participants regardless of their engagement or retention. All intervention content is tailored to TW/MSM with a SUD.

ASK-PrEP is a PrEP navigation intervention with text-messaging support. The navigation component is based on mechanisms of the Reasoned Action Approach (RAA), and the text-messaging support component is based on Social Support Theory (SST). In Session 1, the PrEP navigator uses the Needs and Barriers Assessment (NBA) to identify needs and barriers to PrEP care, including substance use and behavioral health needs; adherence goal(s); and methods to achieve adherence. PrEP (Truvada, Descovy, Cabotegravir) and clinic options are discussed. Per current state-of-the-field recommendations, participants are guided to receive same-day PrEP linkage to their chosen clinic, with the goal of PrEP initiation within the first week of enrollment. In Sessions 2-5, PrEP navigators use the information from the NBA to help the participant overcome barriers to PrEP adherence, and work with participants to address their SUD and need for additional auxiliary services. A shorter version of the NBA (NBA-Lite) is administered at the beginning of Sessions 2-5 as a check-in, and to assess progress through the PrEP Care Continuum; client-centered treatment plans are reviewed and revised as needed. In the ASK-PrEP sessions, client-centered dialogical strategies premised on RAA: 1) identify barriers to PrEP, including substance use; 2) identify participants' readiness to address their SUD and link into other auxiliary needed services; and 3) increase participants' skills and self-efficacy in working with PrEP providers and other social service and treatment facilities. Using a client-centered approach, the PrEP navigator works to link participants into SUD treatment and other ancillary behavioral health and support services, according to their unique barriers, with the ultimate goal of PrEP initiation, adherence, and persistence; services may include mental healthcare, counseling for intimate partner violence, food insecurity, housing instability, hormone therapy. Discussions of PrEP adherence, reductions in substance use and/or substance use treatment, and other behavioral health concerns are discussed throughout the 5 sessions. A key feature of the study is the tailoring of PrEP navigation and text-messaging support to TW/MSM with a SUD.

The text-messaging support component of ASK-PrEP is based in SST. One PrEP support text message is transmitted weekly on Wednesday afternoon between 3:00 - 6:00, participants may choose to have the text messages delivered via cell phone or email. To maintain interest and enthusiasm for the intervention, participants receive TW- or MSM-specific messages, and never receive the same message twice.

Contingency Management is based on behavioral economics. Non-responders are stepped and re-randomized to CM, either in concert with ASK-PrEP, or alone. At the first CM session, a RA provides a 15-minute orientation to the CM procedures, which includes an explanation of the progressive contingency schedule. Thereafter, participants meet with the RA thrice weekly to provide a urine sample. Participants receive a voucher-based escalating reinforcement schedule. Successive urine samples that are nonreactive for the metabolites of their identified SUD will escalate their voucher point value. Each three consecutive nonreactive urine samples will receive bonus voucher points. A reactive urine sample will place the participant at the initial voucher point value; however, a rapid reset procedure allows participants to return to their place in the escalating schedule following three consecutive nonreactive urine samples. Voucher points can be redeemed at any time during the study for goods or services that promote a pro-social and healthy lifestyle.

Participants stepped and re-randomized into ASK-PrEP+CM receive the same ASK-PrEP and CM interventions (described above), but in concert to increase intensity and address both SUD and PrEP initiation, adherence and persistence.

The Standard of Care (SOC) arm provides PrEP education, information, and referrals. Those randomized to the SOC arm will receive an approximate 20-30-minute educational session on PrEP, and will be given a PrEP pamphlet and list of clinics that provide PrEP in Los Angeles County (LAC). The same educational session will be repeated following the 3-month follow-up assessment visit.

ELIGIBILITY:
Inclusion Criteria:

* self-identified transgender woman or MSM
* ≥18 years old
* verified HIV negative
* identified as high risk for HIV based on the Los Angeles County criteria
* SUD (injection and non-injection; excluding cannabis (CUD) only

For those who have already initiated PrEP there is an additional eligibility criterion:

* non-protective prophylaxis defined as missed ≥4 doses of PrEP/week during any week in the previous 30 days
* no PrEP care visits in the past 3 months
* willing to provide informed consent; and
* willing to comply with study requirements.

Should a participant be identified as having kidney or liver dysfunction sufficient to contraindicate PrEP use (creatinine clearance <60 mL/min), that individual will be withdrawn from study participation but may re-screen for eligibility once adequate renal and/or liver function has been established and medically documented (≥60 mL/min).

Exclusion Criteria:

* does not identify as a trans woman or male who has sex with men
* under 18 years of age
* HIV positive status
* not identified as high risk for HIV based on the Los Angeles County criteria
* no verified SUD or only CUD
* if already initiated PrEP: PrEP adherent and PrEP care visits in the past 3 months
* unwilling to provide informed consent
* unwilling to comply with study requirements;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified as trans woman or trans feminine, trans masculine individuals who have a sexual identity of either gay or bisexual and identify as a man who has sex with men.
Enrollment: 152 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Rate of PrEP Persistence | 12 months
  For those who initiate oral-daily PrEP, persistence is defined as a co-occurrence of ≥700fmol/punch and ongoing (i.e., minimum one every 3 months) confirmed PrEP care medical visits. At each time point, those who do not initiate PrEP, fail to attend a PrEP medical care visit in a given quarter, and/or evidence a Dried Blood Spot (DBS) of <700 fmol/punch are coded "non-persistent;" participants who initiate PrEP, attend quarterly medical visits, and evidence a DBS ≥700 fmol/punch will be coded "PrEP persistent." For those who initiate long-acting injectable PrEP, persistence is defined as verified documentation of a Cabotegravir injection every 2 months. Participants that discontinue PrEP due to elimination of their illicit drug use and HIV sexual risk behaviors will be categorized as persistent.
Cost-effectiveness | 12 months
  The primary outcome of the cost-effectiveness analysis is the incremental cost-effectiveness ratio (ICER), which will be calculated as the incremental mean cost of a given intervention relative to an alternative, divided by the incremental mean effectiveness of the two interventions. The primary measure of effectiveness for the economic evaluation will be the quality-adjusted life-year (QALY). The QALY is a measure that combines the health-related quality-of-life (HRQoL) associated with an individual's health state and their time spent in that state. All measures of mean cost and effectiveness will be adjusted for important covariates.
Average Cumulative Days of Substance Use | 12 months
  The primary substance use outcome is cumulative days of the identified illicit substance use measured via timeline follow-back (TLFB), not contraindicated by urine drug screen results. Missing urine drug screens will be treated as positive. Treatment effects will be quantified in terms of the difference in average cumulative days of the identified substance use at 3-, 6-, 9-, and 12-month follow-up visits.

SECONDARY OUTCOMES:
Effects of substances, route of administration, severity of SUD, social and structural determinants of health, and differing individual-level characteristics as moderators. | 12 months
  Longitudinal targeted minimum loss-based estimation (LTMLE) is utilized to estimate subgroup-specific treatment effects based on participant-level characteristics. The magnitude of intervention effects will be compared across relevant subgroups to infer moderation of intervention outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy J Reback, PhD, Principal Investigator — Friends Research Institute, Inc.; Sean M Murphy, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Friends Community Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share IPD.

REFERENCES:
- [Derived] Reback CJ, Landovitz RJ, Benkeser D, Jalali A, Shoptaw S, Li MJ, Mata RP, Ryan D, Jeng PJ, Murphy SM. Protocol for a randomized controlled trial with a stepped care approach, utilizing PrEP navigation with and without contingency management, for transgender women and sexual minority men with a substance use disorder: Assistance Services Knowledge-PrEP (A.S.K.-PrEP). Addict Sci Clin Pract. 2024 Nov 9;19(1):79. doi: 10.1186/s13722-024-00482-6. PMID 39521970